CLINICAL TRIAL: NCT06101862
Title: Team-based Interventional Triage in Acute Coronary Syndrome Based on Non-Invasive Computed Tomography Coronary Angiography - a Randomized Trial
Brief Title: Coronary Computed Tomography Versus Invasive Angiography for Non-ST Elevation Acute Coronary Syndrome
Acronym: TRACTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Niels Thue Olsen, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-23024848
Record Dates: First submitted 2023-09-28; First posted 2023-10-26 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Heart Disease; Non STEMI; Angina Pectoris, Unstable; Coronary Disease; Heart Attack; Acute Myocardial Infarction (AMI); Randomized Controlled Trial; Diagnostic Imaging; Coronary Stenoses; Coronary Artery Disease; Multidetector Computed Tomography; Percutaneous Coronary Intervention
Keywords: Angiography; Computed Tomography; Coronary; Non-STEACS; CCTA; ICA; Randomized; Interventional Triage; TRACTION; Diagnostic imaging; Interventional cardiology; VERDICT; CT; Coronary Angiography; Complications; Coronary CT-team; Ischemic heart disease; Acute myocardial infarction; Non-ST-elevation myocardial infarction (NSTEMI); Unstable angina pectoris; Percutaneous coronary intervention; Coronary artery bypass grafting; PCI; CABG; Diagnostic procedure; Interhospital transfers; Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia; Non-ST Elevated Myocardial Infarction; Angina, Unstable; Coronary Disease; Myocardial Infarction; Coronary Stenosis; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coronary computed tomography angiography + team-based interventional triage (Active Comparator)
  Interventions: Procedure: CCTA; Other: Team-based interventional triage
- Conventional invasive coronary angiography (Other)
  Interventions: Procedure: Conventional ICA

INTERVENTIONS:
Procedure: CCTA — Participants will be examined with CCTA during admission.
  Arms: Coronary computed tomography angiography + team-based interventional triage
Procedure: Conventional ICA — Patients will be examined with conventional standard-of-care ICA.
  Arms: Conventional invasive coronary angiography
Other: Team-based interventional triage — The CCTA will be discussed at a coronary CT-team conference to establish the treatment strategy and provide guidance for any necessary interventional procedure.
  Arms: Coronary computed tomography angiography + team-based interventional triage

SUMMARY:
Coronary computed tomography angiography (CCTA) is a widely accepted initial diagnostic test for individuals suspected of having chronic coronary syndromes. However, there is limited evidence supporting its use in the acute setting. So far, no large-scale randomized trial has examined the performance of CCTA as an alternative to invasive coronary angiography (ICA) in individuals with non-ST-segment elevation myocardial infarction (NSTEACS).

If CCTA were to replace ICA as a routine procedure for individuals with NSTEACS, it could reduce the risk of complications related to ICA, improve patient comfort, expedite decision-making, and reduce healthcare expenses and interhospital transfers.

ELIGIBILITY:
Inclusion criteria:

* Admitted with non-ST-segment elevation myocardial infarction or unstable angina pectoris and an indication for subacute ICA
* Elevated troponin or ischemic electrocardiographic changes
* Written informed consent

Exclusion criteria:

* Instability requiring acute or emergent ICA
* History of percutaneous coronary intervention or coronary artery bypass grafting
* Estimated glomerular filtration rate < 30 mL/min/1.73m2
* Probable type 2 acute myocardial infarction
* Severe valvular heart disease as primary diagnosis or potential need for valve intervention
* History of spontaneous coronary artery dissection
* Expected poor quality of the CCTA
* Prior CCTA or ICA during index admission or within 1 week
* Known allergy to beta-blockers or contrast agent
* Pregnant or nursing
* Previously randomized in this trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2300 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2036-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a combined endpoint of major adverse cardiac events | At 1 year.
  All-cause mortality, non-fatal myocardial infarction, hospitalization with refractory angina, or hospitalization with heart failure.

SECONDARY OUTCOMES:
Number of participants with a the individual composites of the primary outcome | At 1 year.
  All-cause mortality, non-fatal myocardial infarction, hospitalization with refractory angina, or hospitalization with heart failure.
Number of participants with cardiovascular death | At 1 year.
Number of participants with unplanned coronary revascularization | At 1 year.
Health-related Quality of life | At 1 year.
  Measured by EQ-5D-5L
Angina symptom burden | At 1 year.
  Measured by Seattle Angina Questionnaire
Total (cumulative) radiation dosage during index admission | At 1st hospital discharge, an average of 2 days.
Length of index hospitalization | At 1st hospital discharge, an average of 2 days.

CONTACTS AND LOCATIONS:
Locations (6):
- Denmark (6):
  - Herlev and Gentofte Hospital, Copenhagen, Hellerup
  - Bispebjerg Hospital, Bispebjerg
  - Rigshospitalet, Copenhagen
  - Zealand University Hospital, Copenhagen
  - North Zealand Hospital, Hillerød
  - Hvidovre Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request and uploaded to a repository after the trial has been concluded.

REFERENCES:
- [Derived] Sorgaard MH, Kristensen AT, Eskesen K, Kofoed KF, Linde JJ, Kelbaek H, Ottesen M, Neland K, Kragelund C, Bertelsen MLN, Hove JD, Mork G, Kristiansen OP, Engstrom T, Lonborg JT, Kuhl JT, Risom SS, Blanche P, Olsen NT. Coronary computed tomography angiography versus invasive coronary angiography for interventional triage in acute coronary syndrome: Design of the randomized TRACTION trial. Am Heart J. 2025 Dec 6;294:107325. doi: 10.1016/j.ahj.2025.107325. Online ahead of print. PMID 41360328

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-10-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT06101862/SAP_000.pdf